CLINICAL TRIAL: NCT01099761
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ACE-031 (ActRIIB-IgG1) in Subjects With Duchenne Muscular Dystrophy
Brief Title: Study of ACE-031 in Subjects With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on preliminary safety data.
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A031-03
Record Dates: First submitted 2010-04-02; First posted 2010-04-08 (Estimated); Results first posted 2016-10-14 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-09

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ACE-031 0.5 mg/kg q4wk (Experimental)
  Interventions: Biological: ACE-031 0.5 mg/kg q4wk
- ACE-031 1.0 mg/kg q2wk (Experimental)
  Interventions: Biological: ACE-031 1.0 mg/kg q2wk
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ACE-031 0.5 mg/kg q4wk — ACE-031 0.5 mg/kg subcutaneously once every 4 weeks for 12 weeks.
  Arms: ACE-031 0.5 mg/kg q4wk
Biological: ACE-031 1.0 mg/kg q2wk — ACE-031 1.0 mg/kg subcutaneously once every 2 weeks for 12 weeks.
  Arms: ACE-031 1.0 mg/kg q2wk
Other: Placebo — Matching volume placebo subcutaneously every 2 or 4 weeks for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if ACE-031 is safe and well-tolerated in boys with Duchenne Muscular Dystrophy (DMD) and to select the optimal doses of ACE-031 in terms of safety and pharmacodynamic (PD) activity for designing future studies. [Note: This study was terminated based on safety data]

DETAILED DESCRIPTION:
ACE-031, a soluble form of the human activin receptor type IIB, was administered once every 2 to 4 weeks by subcutaneous (SC) injection to boys with DMD. Dose levels and regimens for this multiple-dose study were based on data from the initial clinical studies in healthy subjects in which doses of 0.02 to 3 mg/kg SC were evaluated. A total of 24 subjects were enrolled into the study; 18 received ACE-031 and 6 placebo. All subjects were treated for a period of 12 weeks.The pharmacodynamic effects of ACE-031 treatment were assessed by a battery of motor function test that included the 6-Minute Walk Test, the 10-Minute Walk/Run Test, the 4-Stair Climb Test and the Gower Maneuver (GW). Muscle strength was assessed by hand-held myometry and fixed system testing. Body composition (i.e., spine BMD, lean mass, and fat mass) was assessed by whole body and lumbar spine DXA scans. Pulmonary function was assessed by forced vital capacity (FVC), maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP). ACE-031 safety was evaluated through observation of the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed
* Ambulant
* Corticosteroid therapy for at least one year prior to study day 1 and on a stable dose and schedule for at least 6 months prior to study day 1
* Evidence of muscle weakness by clinical assessment

Exclusion Criteria:

* Any previous treatment with another investigational product within 6 months prior to study day 1
* Any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease that is not related to DMD
* Inability to perform a whole body dual x-ray absorptiometry (DXA) scan

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Acceleron Investigative Site, Calgary, Alberta
  - Acceleron Investigative Site, Vancouver, British Columbia
  - Acceleron Investigative Site, Hamilton, Ontario
  - Acceleron Investigative Site, London, Ontario
  - Acceleron Investigative Site, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
Abstract summarizing trial data has been published online in Muscle & Nerve 23-Dec-2016 https://www.ncbi.nlm.nih.gov/pubmed/27462804 The Sponor currently has no plans to make IPD available for a number of reasons; (i) the study was terminated by the Sponsor prematurely based upon concerns for potential adverse drug reactions following long-term use, which were identified in chronic toxicity studies in animals, (ii) the study population was one with a rare disease, in a groups of subjects with a relatively narrow age range, across a small number of study sites. The Sponsor believes that these factors, taken together, make patient anonymity a significant challenge.

RESULTS

PARTICIPANT FLOW:
Groups:
- ACE-031 ACE-03 2.5 mg/kg q4wk: ACE-031 2.5 mg/kg q4wk: ACE-031 2.5 mg/kg subcutaneously once every 4 weeks for 12 weeks.
Period: Overall Study
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | ACE-031 ACE-03 2.5 mg/kg q4wk | Placebo
Started | 9 | 9 | 0 (Study terminated prior to enrolling cohort 3) | 6
Completed | 9 | 9 | 0 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | ACE-031 ACE-03 2.5 mg/kg q4wk | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 0 | 6 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 |  | 6 | 24
  Between 18 and 65 years | 0 | 0 |  | 0 | 0
  >=65 years | 0 | 0 |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 |  | 0 | 0
  Male | 9 | 9 |  | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0 | 0
  Not Hispanic or Latino | 9 | 9 |  | 6 | 24
  Unknown or Not Reported | 0 | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 9 |  | 6 | 24
Able to ambulate 10 meters in < 12 seconds [Number; unit: participants] | 9 | 9 |  | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Reactions.
Description: Number of subjects in each cohort with a treatment-emergent adverse event considered at least possibly related to study drug
Time Frame: From treatment initiation to End-of-Study Visit, approximately 24 weeks later
Measure: Number; unit: Number of subjects
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
Number of subjects | 1 | 6 | 0

2. Primary Outcome: Number of Subjects With Clinical Laboratory Adverse Reactions.
Description: Number of subjects in each cohort with treatment-emergent adverse laboratory values judged to be at least possibly related to study drug
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Number; unit: Number of subjects
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
Number of subjects | 0 | 0 | 0

3. Secondary Outcome: Percent Change in Total Lean Body Mass by DXA Scan.
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Error); unit: percentage change in lean body mass
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
percentage change in lean body mass | 3.6 (1.3) | 4.1 (1.5) | 2.6 (1.8)
Statistical Analysis 1: Comparison: ACE-031 0.5 mg/kg q4wk; Test type: Superiority or Other; p = 0.023, ANCOVA
Statistical Analysis 2: Comparison: ACE-031 1.0 mg/kg q2wk; Test type: Superiority or Other; p = 0.012, ANCOVA
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; p = 0.435, ANCOVA

4. Secondary Outcome: Percent Change in Lumbar Spine Bone Mineral Density by DXA Scan.
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
percentage change from baseline | 1.6 (1.8) | 4.4 (1.5) | 0.3 (4.4)
Statistical Analysis 1: Comparison: ACE-031 1.0 mg/kg q2wk; Test type: Superiority or Other; p = 0.039, ANCOVA

5. Secondary Outcome: Percent Change in Muscle Strength Score by Hand-held Myometry.
Description: Manual Muscle Testing (MMT) is a procedure to measure the function and strength of individual muscles and muscle groups. Hand-held myometry, using a device known as a dynamometer, is one method used for MMT. The dynamometer is held against the patient's limb by the examiner and the patient is asked to resist the force applied by the examiner. The dynamometer measures the force applied by the patient, providing a quantitative and objective assessment of strength of the particular muscle or muscle group. The effectiveness of a therapeutic intervention on muscle strength, as measured by hand-held myometry, can be assessed by comparing post-treatment to pre-treatment (baseline) measurements.
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
percentage change from baseline
  Elbow extension (kg) | 0.3 (3.2) | 0.1 (2.3) | -0.1 (2.1)
  Elbow flexion (kg) | -0.4 (3.4) | -0.7 (2.6) | 0.3 (3.1)
  Knee extension (kg) | -3.6 (4.4) | -3.3 (4.4) | -3.7 (5.0)
  Knee flexion (kg) | -2.2 (3.1) | -1.9 (4.1) | -1.2 (3.9)

6. Secondary Outcome: Change in Distance Traveled in 6 Minutes (Standardized 6-Minute-Walk Test).
Description: Change in distance traveled in 6 minutes (standardized 6-Minute-Walk Test); stratified by baseline age (<10 years vs. >=10 years)
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Deviation); unit: change (m) in 6MWT from baseline
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
change (m) in 6MWT from baseline
  <10 years of age at baseline | 43.8 (61.5) | 2.5 (35.6) | 5.2 (23.6)
  >=10 years of age at baseline | 4.5 (37.6) | -3.2 (35.5) | -47.6 (34.5)

7. Secondary Outcome: Change From Baseline in Time to Travel 10 Meters (Standardized 10-Meter-Walk/Run Test).
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Deviation); unit: Change (sec) in 10MWT from baseline
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
Change (sec) in 10MWT from baseline | 0.7 (0.9) | 0.7 (0.9) | 1.0 (0.8)

8. Secondary Outcome: Change in Pulmonary Function Tests (FVC)
Description: Forced Vital Capacity (FVC); 1 of 3 separate tests employed to assess pulmonary function in this study
Time Frame: Baseline to End-of-Study Visit, approximately 24 weeks later.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
Liters | 0.1 (0.2) | 0.1 (0.1) | 0.1 (0.2)

9. Secondary Outcome: Change in Pulmonary Function Test (MIP)
Description: Maximum Inspiratory Pressure (MIP); 2 of 3 separate tests employed to assess pulmonary function in this study
Time Frame: Baseline to End-of-Study Visit. approximately 24 weeks
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
cm H2O | 17.2 (17.2) | 8.7 (7.6) | 8.8 (22.1)

10. Secondary Outcome: Change in Pulmonary Function Test (MEP)
Description: Maximum Expiratory Pressure (MEP); 3 of 3 separate tests employed to assess pulmonary function in this study
Time Frame: Baseline to End-of-Stuidy Visit, approximately 24 weeks
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | Placebo
Number analyzed (Participants) | 9 | 9 | 6
cm H2O | 11.9 (12.5) | 0.8 (3.9) | 5.8 (12.1)

ADVERSE EVENTS:
Time Frame: 24 weeks (12 weeks treatment period + 12 weeks follow up)
Arm/Group | ACE-031 0.5 mg/kg q4wk | ACE-031 1.0 mg/kg q2wk | ACE-031 ACE-03 2.5 mg/kg q4wk | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/0 | 0/6
Other Adverse Events (participants affected / at risk) | 3/9 | 6/9 | 0/0 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACE-031 0.5 mg/kg q4wk (N=9) | ACE-031 1.0 mg/kg q2wk (N=9) | ACE-031 ACE-03 2.5 mg/kg q4wk (N=0) | Placebo (N=6)
Injection site erythema (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 3
epistaxis (Vascular disorders) | 1 | 5 | 0 | 0
telangiectasia (Vascular disorders) | 0 | 5 | 0 | 0
headache (General disorders) | 1 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No